CLINICAL TRIAL: NCT01145872
Title: The Effects and Mechanisms of MBCT on Depressive Symptoms and Depression Relapse
Brief Title: The Effects and Mechanisms of Mindfulness Based Cognitive Therapy (MBCT) on Depressive Symptoms and Depression Relapse
Acronym: MBCT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Denver (Other)
Collaborators: Stanford University (Other); University of Colorado, Boulder (Other)
Responsible Party: Principal Investigator, Amanda Shallcross, Post-Doctoral Researcher, University of Denver
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: F32AT004879-01A2 (NIH)
Record Dates: First submitted 2010-06-16; First posted 2010-06-17 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-12

CONDITIONS: Major Depressive Disorder; Recurrent
Keywords: Mindfulness; clinical trial; intervention; prevention
MeSH Terms: conditions — Depressive Disorder, Major; Recurrence | interventions — Mindfulness-Based Cognitive Therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mindfulness Based Cognitive Therapy (Experimental)
  Interventions: Behavioral: Mindfulness Based Cognitive Therapy
- Health Enhancement Program (Active Comparator)
  Interventions: Behavioral: Health Enhancement Program

INTERVENTIONS:
Behavioral: Mindfulness Based Cognitive Therapy
  Arms: Mindfulness Based Cognitive Therapy
Behavioral: Health Enhancement Program
  Arms: Health Enhancement Program

SUMMARY:
This research proposal is intended to elucidate the efficacy and mechanisms underlying Mindfulness Based Cognitive Therapy (MBCT) in a population in remission from recurrent Major Depressive Disorder (MDD). The first objective of the study is to replicate previous studies' findings of MBCT's effects on decreasing depressive symptoms and depression relapse rates. However, this proposal aims to make a novel contribution to the literature by using a randomized, controlled design, and comparing the effects of MBCT to an active control condition (ACC). The use of a well-designed ACC will enable us to control for confounding variables such as social support and expected outcomes, thus allowing us to determine whether elements specific to MBCT lead to its salutary effects (Aim 1). Previous MBCT studies have largely relied on self-report measurement methodologies, limiting valid conclusions about the nature of MBCT. Further, few studies have examined the mechanisms underlying effects of MBCT on depressive symptoms and relapse. Theoretical considerations and preliminary empirical evidence suggest emotional, physiological, and cognitive functioning to be promising mechanisms of MBCT. Therefore, the investigators propose to assess each of these potential mechanisms of MBCT using self-report, autonomic physiological, and reaction time tasks (Aim 2). Collectively, these aims are expected to strengthen the evidence base for MBCT while cultivating a scientific model for its effects and mechanisms on decreasing depressive symptoms and depression relapse rates.

ELIGIBILITY:
Inclusion Criteria:

* must comprehend English well
* be 18-55 years of age
* meet enhanced DSM-IV criteria for remission of MDD, recurrent and have a history of three or more previous episodes of DSM-IV major depression in the absence of a history of mania or hypomania
* at least one of those episodes was within the past two years
* participant must be in remission and if on antidepressant medication (ADM), they must be on a stable dose with no change in type or amount for past 12 weeks or participants must be off ADM at T1 for at least the preceding 12 weeks
* have, at screening assessment, residual depressive symptoms indicated by a Beck Depression Inventory-II (BDI-II;[72]) score between 6-19.

Exclusion Criteria:

* bipolar disorder
* schizophrenia or borderline personality disorder
* current suicidal thoughts and/or suicide attempt in last two months
* current anxiety disorder if it constitutes the predominant aspect of the clinical presentation and requires primary treatment not offered in the project
* substance abuse or dependence within last three months
* dementia or subnormal intellectual potential
* current obsessive-compulsive disorder
* current eating disorder
* history of previous mindfulness training or more than eight lifetime sessions of CBT
* current use of psychotherapy or counseling

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 92 (Actual)
Dates: Start 2010-07; Primary Completion 2012-05 (Actual); Study Completion 2013-04 (Actual)

PRIMARY OUTCOMES:
Depression Relapse | 1 year

SECONDARY OUTCOMES:
Depressive Symptoms | 1 Year

CONTACTS AND LOCATIONS:
Locations (1):
- University of Denver, Denver, Colorado, United States